CLINICAL TRIAL: NCT06005155
Title: Lithium Versus Anticonvulsants and the Risk of Physical Disorders - Results From a Comprehensive Long-term Nation-wide Population-based Study Emulating a Randomised Trial
Brief Title: Lithium Versus Anticonvulsants and the Risk of Physical Disorders
Status: Completed | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Lithium versus anticonvulsants
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Disorder
Keywords: Lithium; Lamotrigerne; Valproate; Physical disorders
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Valproic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lithium — Sustained long-term exposure
  Other Names: Lamotrigene; Valproate

SUMMARY:
Nationwide population-based register linkage study covering the entire 5.9 million inhabitants in Denmark systematically investigating the associations between sustained long-term use of lithium versus lamotrigine and valproate, and the risk of a range of physical disorders emulating a randomized trial.

DETAILED DESCRIPTION:
The study includes two cohorts. Cohort 1: all 12.607 patients with a diagnosis of bipolar disorder (ICD-10 code: DF30-31.9) who subsequently were exposed to either lithium, lamotrigine or valproate between 1997 and 2021. Cohort 2: as Cohort 1, but regardless of prior diagnosis of bipolar disorder (N= 156.678).

Main analyses considered a patient exposed to a drug 92 days after a prescription and a 10-year follow-up and 4 sensitivity analyses considered a patient exposed to a drug for 60 and 180 days after a prescription, respectively, and with 5- and 15-years follow-up, respectively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bipolar disorder and subsequent exposure to either lithium, lamotrigine or valproate

Exclusion Criteria:

* None

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nationwide population-based register linkage study covering the entire 5.9 million inhabitants in Denmark and two cohorts. Cohort 1: all 12.607 patients with a diagnosis of bipolar disorder (ICD-10 code: DF30-31.9) who subsequently were exposed to either lithium, lamotrigine or valproate between 1997 and 2021. Cohort 2: as Cohort 1, but regardless of prior diagnosis of bipolar disorder (N= 156.678).
Sampling Method: Non-Probability Sample
Enrollment: 169285 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incident stroke (separately for intracerebral hemorrhage and cerebral infarction) | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Arteriosclerosis | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Angina pectoris | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Myocardial infarction | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Diabetes mellitus (separately for type 1 diabetes and type 2 diabetes) | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Myxoedema | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Osteoporosis | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Dementia (separately for Alzheimer's disease and other dementia) | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Parkinson's disease | 1997 to 2021
  Diagnosis in the Danish National Hospital Register
Chronic kidney disease (definite chronic kidney disease and possible Chronic kidney disease) | 1997 to 2021
  Diagnosis in the Danish National Hospital Register

CONTACTS AND LOCATIONS:
Overall Officials: Lars V Kessing, Professor, Principal Investigator — Psychiatric Center Copenhagen
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark